CLINICAL TRIAL: NCT01248481
Title: Combined Use of a Basal Insulin and Glucobay For Reducing PPG to End Diabetes Progress
Brief Title: GlucoFriend-evaluation the Effectiveness of Glucobay When Combined With a Basal Insulin
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Country Medical Director, Bayer Healthcare AG
Other Study IDs: 15316; GB1010KR (Other: Company Internal)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus
Keywords: Acarbose/Glucobay®; Basal insulin; PPG (Postprandial Glycaemia)
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)

INTERVENTIONS:
Drug: Acarbose (Glucobay, BAYG5421) — Adult female and male patients are scheduled to be treated with acarbose will be enrolled after the therapy decision has been made. Physicians should consult the full prescribing information for Glucobay® before enrolling patients and familiarize themselves with the safety information in the product package label.

SUMMARY:
To evaluate the effectiveness of Glucobay when combined with a basal insulin under daily-life treatment conditions in a large sample of Korean patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 18 years
* Diagnosed of type 2 diabetes for at least 6 months prior to enrollment
* Patients treated with stable dose of a basal insulin (insulin glargine or insulin detemir) at least 2 months
* HbA1C≥7.5 and ≤10.0%

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DM in korea
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2010-09; Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | After 20 weeks

SECONDARY OUTCOMES:
Duration and dose of acarbose treatment | After 20 weeks
Postprandial Blood Glucose | After 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea